CLINICAL TRIAL: NCT01845558
Title: Effects of Wobenzym® Plus in Healthy, Sportive People After Eccentric Exercise - a Randomized, Two-stage, Double-blind, Placebo-controlled Cross-over Trial
Brief Title: Effects of Wobenzym® Plus in Healthy, Sportive People After Eccentric Exercise
Acronym: 2012-005003-40
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mucos Pharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTS651/12; 2012-005003-40 (EudraCT Number)
Record Dates: First submitted 2013-04-23; First posted 2013-05-03 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Muscle Injury; Muscle Soreness; Exercise Induced Muscle Damage
Keywords: Muscle soreness; Exercise induced muscle damage; Inflammation; Proteolytic enzymes; Muscle strength Dynamometer
MeSH Terms: conditions — Myalgia; Inflammation | interventions — Wobenzym

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wobenzym® plus (Experimental): Treatment with the licenced drug Wobenzym® plus (3x4 Capsules/ day)
  Interventions: Drug: Wobenzym® plus
- Placebo equates Wobenzym® plus but without active ingredients (Placebo Comparator): 3x4 capsules/ day
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Wobenzym® plus
  Arms: Wobenzym® plus
Other: Placebo
  Arms: Placebo equates Wobenzym® plus but without active ingredients

SUMMARY:
The aim of the current study is to investigate the therapeutic effect and especially the mode of action of Wobenzym® plus, an anti-inflammatory drug containing proteolytic enzymes, on exercise induced muscle damage (eiMD) and recovery time in male amateur sportsmen with medium proficiency level compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations
* Subject is in good physical and mental health as established by medical history, physical examination, electrocardiogram, vital signs, results of biochemistry, haematology
* Not anticipating any planned changes in lifestyle regarding activity and nutrition for the duration of the study
* Non smoker
* Men with strength training experience
* Age: 20-50 years
* BMI ≥20 kg/m2 and ≤ 32 kg/m2
* medium concentric strength ability (150-300 Nm)

Exclusion Criteria:

* Relevant history or presence of any medical disorder, potentially interfering with this trial (e.g. volunteers having experienced any cardiovascular events such as infarction, angina, surgical endocoronary intervention, stroke or volunteers suffering from diabetes as well as acute or chronic injury of the musculoskeletal system, e.g. cruciate ligament rupture.
* No intake of anti-inflammatory medication/ food supplements or intake of medications that directly affect parameters of muscle function or performance within 4 weeks prior to visit 1 or during the trial
* Subjects not willing to abstain from intake of analgesic medication 24 hours prior to and during visit 1 and 2.
* For this trial clinically relevant abnormal laboratory, vital signs or physical findings at screening
* Known hypersensitivity to the study preparation or to single ingredients (e.g. Lactose intolerance)
* Drug, alcohol and/or medication abuse
* Known HIV-infection
* Known acute or chronic hepatitis B and C infection
* Participation in another clinical trial within the last 4 weeks and concurrent participation in another clinical trial
* Blood donation within 4 weeks prior to trial start (visit 1) or during trial.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Reduction of maximal concentric strength, movement induced pain and pressure induced pain combined in a multidimensional (composite outcome)model giving information about the change induced by the stress test | immediately before, 24h post, 48h post
  Multidimensional approach for recovery and acute phase after eccentric stress test. Will be assessed at different time points before and after an excentric stress test and the reduction of these parameters under treatment will be calculated.

SECONDARY OUTCOMES:
Maximal concentric strength (Nm) before and after the stress test | immediately before, 0h, 3h, 6h, 24h, 48h, 72h
  Reduction of strength induced by the excentric stress test
Pressure induced pain | immediately before, 0h, 3h, 6h, 24h, 48h, 72h
  Pain induced by the stress test rated via Algometry kg/cm*cm induced by standardised pressure
Blood routine parameters | immediately before, 0h, 3h, 6h, 24h, 48h, 72h
  Blood routine parameters (differentiated haemogram; blood lipids; glucose; kreatinin) as safety parameters
blood pressure | immediately before, 24h, 48h, 72h
  Blood pressure and heart rate as safety parameter
Movement induced pain | immediately before, 0h, 3h, 6h, 24h, 48h, 72h post
  Pain induced by a standardised movement and rated by the volunteer via VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Pabst, Dr. med, Principal Investigator — PWC GmbH
Locations (1):
- Sportschule FFb Puch GmbH, Fürstenfeldbruck, Germany